CLINICAL TRIAL: NCT06019637
Title: A Long-term Safety Study in Brazilian Patients With a Confirmed Diagnosis of Spinal Muscular Atrophy (SMA) Treated With Onasemnogene Abeparvovec (Zolgensma®) - ARISER Study
Brief Title: A Long-term Safety Study in Brazilian Patients With a Diagnosis of Spinal Muscular Atrophy Treated With Zolgensma
Acronym: ARISER
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COAV101ABR01
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Spinal Muscular Atrophies
Keywords: Spinal Muscular Atrophies;; Onasemnogene Abeparvovec;; Brazil;; NIS
MeSH Terms: interventions — Zolgensma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Spinal Muscular Atrophy Patients: Brazilian pediatric patients with a confirmed diagnosis of Spinal Muscular Atrophy treated with Onasemnogene Abeparvovec
  Interventions: Other: Onasemnogene Abeparvovec

INTERVENTIONS:
Other: Onasemnogene Abeparvovec — Retrospective and prospective observational study. There is no treatment allocation.
  Other Names: Zolgensma

SUMMARY:
A long-term safety study in Brazilian patients with a confirmed diagnosis of Spinal Muscular Atrophy (SMA) treated with Onasemnogene Abeparvovec (Zolgensma®)

DETAILED DESCRIPTION:
This study is a non-interventional Post Authorization Safety Study (PASS) to evaluate long-term, real-world safety data of Brazilian pediatric patients diagnosed with SMA and treated with Onasemnogene Abeparvovec (Zolgensma®) for up to 15 years after the treatment. This study will support the benefit-risk assessment of Onasemnogene Abeparvovec in the approved indications and may also allow for detection of new safety signals and provide further guidance on the management of safety risks associated with Onasemnogene Abeparvovec to patients/caregivers, health care providers (HCPs) and treating physicians, as required by Brazilian Health Authority ANVISA as a conditional measure for granting Zolgensma®'s authorization.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent or legal guardian has provided signed eICF.
* Subject with SMA, genetically confirmed: with a bi-allelic mutation in the SMN1 gene, and a clinical diagnosis of SMA Type 1 or up to 3 copies of the SMN2 gene.
* Subject treated* with Onasemnogene Abeparvovec (Zolgensma®) prior to enrolling in this study.

Subjects treated with nusinersen or risdiplam prior to Onasemnogene Abeparvovec (Zolgensma®) can be enrolled if currently not receiving it.

*Subjects can be enrolled in this study on the day treated with Onasemnogene Abeparvovec (Zolgensma®) or if prior medical history is available to complete all assessments retrospectively, in accordance with local ethical requirements.

* Subject and parent/guardian are willing and able to comply with the phone contacts through the course of the study

Exclusion Criteria:

* Patients currently enrolled in any interventional clinical trial** other than the phase IV OFELIA trial will be excluded from the study.

  * Subjects who were enrolled in a clinical trial (independently of the disease indication and interventional treatment) but are not currently enrolled, can be included in this study.

During the follow-up, subjects who enroll any clinical trial with pharmacological intervention will discontinue from this study.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of approximately 50 Brazilian pediatric patients with SMA who were treated with Onasemnogene Abeparvovec (Zolgensma®) in the commercial setting, the closed MAP, or the phase IV OFELIA trial. Patients will be recruited in up to 3 centers in Brazil, over one year of recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2038-09-30 (Estimated); Study Completion 2038-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent SAEs | Up to 5 years
  Incidence and severity of treatment-emergent Serious AEs (SAEs)

SECONDARY OUTCOMES:
Number of patients who experience at least one AESI and number of patients by AESI | Up to 15 years
  Adverse Event of Special Interest: thrombocytopenia, hepatotoxicity, thrombotic microangiopathy (TMA), dorsal root ganglia toxicity, cardiac AEs, new malignancies, new incidence of neurologic, autoimmune, and hematologic disorder
Number of patients who have survived and have not required permanent ventilatory assistance | Up to 15 years
  Evaluation of permanent ventilatory assistance, defined as requiring invasive ventilation(tracheostomy), or respiratory assistance for 16 or more hours per day (including non-invasiveventilatory support) continuously for 14 or more days in the absence of an acute reversible illness,excluding perioperative ventilation.
Time until death or the need for permanent ventilatory assistance | Up to 15 years
  Evaluation of permanent ventilatory assistance, defined as requiring invasive ventilation(tracheostomy), or respiratory assistance for 16 or more hours per day (including non-invasiveventilatory support) continuously for 14 or more days in the absence of an acute reversible illness,excluding perioperative ventilation.
Number of patients who achieve each Developmental Motor Milestone | Up to 15 years
  Evaluation of WHO Developmental Milestones: sitting without support, hands, and knees crawling, standing with assistance, walking with assistance, standing alone, and walking alone.
Number of patients who achieve each WHO Developmental Milestone within age percentiles | Up to 15 years
  Evaluation of WHO Developmental Milestones: sitting without support, hands, and knees crawling, standing with assistance, walking with assistance, standing alone, and walking alone.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Brazil (2):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No